CLINICAL TRIAL: NCT05303831
Title: Pattern of Disease and Determinants of Clinical Outcomes Among ICU Patients on Mechanical Ventilator in Southern Ethiopia: A Multi-center Prospective Cohort Study
Brief Title: Pattern of Disease and Determinants of Clinical Outcomes Among ICU Patients
Acronym: PDCO
Status: Completed | Type: Observational
Sponsor: Dilla University (Other)
Responsible Party: Principal Investigator, Semagn Mekonnen, Assistant professor, thematic research leader, Dilla University
Other Study IDs: duirb/001/21-08
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Clinical Outcomes
MeSH Terms: interventions — Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mechanical ventilator — patients on a mechanical ventilators in ICU will be followed for 28-days for clinical outcomes

SUMMARY:
The global mortality rate of patients on MV is very high which is varied with the income level of the country, duration of a mechanical ventilator, the pattern of disease, ICU staff profile, availability of medical supplies. All Studies conducted so far in Sub-Saharan Africa including Ethiopia among ICU patients primarily focused on the pattern of admission, the incidence of mortality, and its determinants. However, the body of evidence on the pattern of disease, the incidence of MV, and determinants of mortality among patients on MV is still uncertain and a topic of debate nationally as well as locally.

Therefore, A multicenter prospective cohort study is planned to be carried out in Southern Ethiopia Teaching and referral hospital ICUs.

DETAILED DESCRIPTION:
Introduction: The global mortality rate of patients on MV is very high which is varied with the income level of the country, duration of a mechanical ventilator, the pattern of disease, ICU staff profile, availability of medical supplies. All Studies conducted so far in Sub-Saharan Africa including Ethiopia among ICU patients primarily focused on the pattern of admission, the incidence of mortality, and its determinants. However, the body of evidence on the pattern of disease, the incidence of MV, and determinants of mortality among patients on MV is still uncertain and a topic of debate nationally as well as locally.

Objective: The general objective of the study is to investigate the pattern of disease and determinants of mortality among ICU patients on Mechanical ventilators in Southern Ethiopia from April 2021 to September 2022.

Methods: After obtaining Ethical clearance from Research Ethics Committee (IRB), a multi-center cohort study will be conducted in three teaching and referral hospitals in Southern Ethiopia; namely, Hawassa university referral hospital (HURH), Dilla University referral hospital (DURH), and Wolaita Sodo referral hospital (WURH) from March 2021, to September 2022. Four Hundred Forty-four consecutive Adult patients who will be on a mechanical ventilator in ICU fulfilling the inclusion criteria and will be followed for 28-days to assess the pattern of disease, survival status and determinants of mortality will be included. Data will be entered into Statistical Package for Social Sciences version 22 for analysis. Descriptive statistics will be run to see the overall distribution of the study subjects concerning the variables under study. Chi-square test and odds ratio will be used to determine the association between hypothesized independent and dependent variables. Multivariate analysis will be conducted to control possible confounders and identify independent predictors of length of ICU stay and 28- days mortality. Survival analysis and Cox regression will be done to estimate the probability of dying within 28 days and time to wean from a mechanical ventilator.

ELIGIBILITY:
Inclusion Criteria: All Adult patients greater than 12 years old and who are on Mechanical ventilators in DURH, Wolaita Sodo University Hospital, and Hawassa University specialized hospital ICUs and staying in ICU for more than 24hrs of Admission

Exclusion Criteria:

* Patients admitted to ICU on re-admission and patients with no attendants will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Adult patients who are on Mechanical ventilator in Dilla University referral hospital, Wolaita Sodo University Hospital, and Hawassa University specialized Hospital ICUs during the study period
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of mortality | 28-days
  The incidence of mortality of patients in the ICU who are on Mechanical ventilator during 28-days follow up
time to death | 28-days
  The time with which patients die during follow up

SECONDARY OUTCOMES:
time to wean from the MV | 28-days
  This refers to the time when patients weaned from the MV
time to develop adverse events | 28-days
  The time with which patients develop complications during follow up such as cardiac arrest, ventilator associated Pneumonia etc.
Incidence of prolonged ventilation | 28-days
  This study intends to investigate how many of patients are on mechanical ventilator for prolonged period during follow up as per the criteria of prolonged MV

CONTACTS AND LOCATIONS:
Locations (1):
- Dilla University, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Abate SM, Basu B, Jemal B, Ahmed S, Mantefardo B, Taye T. Pattern of disease and determinants of mortality among ICU patients on mechanical ventilator in Sub-Saharan Africa: a multilevel analysis. Crit Care. 2023 Jan 24;27(1):37. doi: 10.1186/s13054-023-04316-w. PMID 36694238